CLINICAL TRIAL: NCT04812977
Title: Comparison of Intravitreal Bevacizumab and Triamcinolone Acetonide With Intravitreal Bevacizumab Alone in Macular Edema Secondary to Central Retinal Vein Occlusion
Brief Title: Comparison of Intravitreal Anti-VEGF Versus Combination Therapy in Central Retinal Vein Occlusion
Acronym: CRVO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hayatabad Medical Complex (Other Government)
Responsible Party: Principal Investigator, Yousaf Jamal Mahsood, Dr., Hayatabad Medical Complex
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 094/HEC/PICO/18
Record Dates: First submitted 2021-03-20; First posted 2021-03-24 (Actual); Results first posted 2022-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-04

CONDITIONS: Central Retinal Vein Occlusion With Macular Edema
Keywords: central retinal vein occlusion; macular edema; intravitreal bevacizumab
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): A single injection of triamcinolone acetonide (Kenacort-AⓇ). (2mg/0.05ml) and intravitreal bevacizumab (Avastin®) (1.25mg/0.05ml) was given at the start of the treatment whereas intravitreal bevacizumab (1.25mg/0.05ml) was repeated monthly for 3 months.
  Interventions: Drug: Group A
- Group B (Active Comparator): Intravitreal bevacizumab (1.25mg/0.05ml) was repeated monthly for 3 months.
  Interventions: Drug: Group A

INTERVENTIONS:
Drug: Group A — Combination of intravitreal triamcinolone acetonide (Kenacort-AⓇ) (2mg/0.05ml) and intravitreal bevacizumab (Avastin®) (1.25mg/0.05ml)

SUMMARY:
To compare the effect of intravitreal-Bevacizumab and Triamcinolone with intravitreal-Bevacizumab alone on visual acuity and central foveal thickness in patients with macular edema secondary to central retinal vein occlusion.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of either gender, age 40-80 years, having macular edema secondary to CRVO, Best-corrected visual acuity (BCVA) of less than or equal to 0.3 on Log MAR chart (Snellen equivalent of 6/12), Central foveal thickness CFT greater than or equal to 250 microns on Heidelberg Spectralis Spectral Domain Optical coherence tomography (SD-OCT) and clinical diagnosis of CRVO.

Exclusion Criteria:

* previously received laser treatment and/or intravitreal injection of any Anti-VEGF agent, having one eye, diagnosed case of glaucoma, family history of glaucoma, young patient, and anyone who has received any treatment for CRVO before presenting to us.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-06-10 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2018-12-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hayatabad Medical Complex, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yoshizawa C, Saito W, Kase M, Ishida S. Clinical Features of Central Retinal Vein Occlusion With Inflammatory Etiology. Asia Pac J Ophthalmol (Phila). 2012 Sep-Oct;1(5):270-6. doi: 10.1097/APO.0b013e318266de04. PMID 26107597
- [Background] Lazic R, Boras I, Vlasic M, Gabric N, Tomic Z. Anti-VEGF in treatment of central retinal vein occlusion. Coll Antropol. 2010 Apr;34 Suppl 2:69-72. PMID 21305727

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All enrolled participants completed the study.
Period: Overall Study
Arm/Group | Group A | Group B
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.93 (4.38) | 60.73 (3.67) | 60.83 (4.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 05 | 08 | 13
  Male | 10 | 07 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Pakistan | 15 | 15 | 30
Visual acuity [Mean (Standard Deviation); unit: logMAR units] | 0.87 (0.09) | 0.88 (0.1) | 0.87 (0.09)
central foveal thickness [Mean (Standard Deviation); unit: microns] | 673.67 (38.33) | 674.07 (36.32) | 673.87 (37.33)

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: Change in visual acuity
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: logMAR units
Groups:
- Combination Group: A single injection of triamcinolone acetonide (Kenacort-AⓇ). (2mg/0.05ml) and intravitreal bevacizumab (Avastin®) (1.25mg/0.05ml) was given at the start of the treatment whereas intravitreal bevacizumab (1.25mg/0.05ml) was repeated monthly for 3 months
- Standard Group: group B received IVB (1.25mg/0.05ml) alone
Arm/Group | Combination Group | Standard Group
Number analyzed (Participants) | 15 | 15
logMAR units | 0.32 (0.06) | 0.44 (0.06)

2. Secondary Outcome: Central Foveal Thickness
Description: change in central foveal thickness
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Combination Group | Standard Group
Number analyzed (Participants) | 15 | 15
microns | 264.4 (16.73) | 271.01 (20.14)

ADVERSE EVENTS:
Time Frame: 6 months.
Arm/Group | Combination Group | Standard Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-07): https://cdn.clinicaltrials.gov/large-docs/77/NCT04812977/Prot_SAP_000.pdf